

**Boehringer Ingelheim** 

# STATISTICAL ANALYSIS PLAN

## **Study Title**

A regulatory required non-interventional study to monitor the safety and effectiveness of Ofev (Nintedanib 150mg/100mg BID) in Korean patients

**Protocol No./Version** 

1199-0417/3.1

**Sponsor** 

Version No.

1.0



## SIGNATURE PAGE

| Prepared by: | | |
|------------------------------------|-----------|--------------------|
| /Biostatistician Name/ Role | Signature | Date (DD-MMM-YYYY) |
| Reviewed/Approved by: | | |
| /Senior Biostatistician Name/ Role | Signature | Date (DD-MMM-YYYY) |



| Approved by Sponsor: | | |
|----------------------|-----------|--------------------|
| /NIS | | |
| Name/ Role | Signature | Date (DD-MMM-YYYY) |



# **VERSION INFORMATION** (DOCUMENT REVISION HISTORY)

| Version | Date | Prepared by | Details |
|---------|-------------|-------------|---------------|
| 1.0 | 04-MAY-2022 | | First Version |
| 150 | | | |



## ABBREVIATION

| Term | Definition |
|---|---|
| ADR | Adverse drug reaction |
| AE | Adverse events |
| AESI | Adverse events of special interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| DB | Database |
| FVC | Forced vital capacity |
| HRCT | High resolution computed tomography |
| IPF | Idiopathic pulmonary fibrosis |
| MFDS | Ministry of food and drug safety |
| PF-ILD | Progressive fibrosing interstitial lung disease |
| PT | Preferred term |
| SADR | Serious adverse drug reaction |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Supporting document |
| SOC | System organ class |
| SOP | Standard operating procedure |
| SS | Safety set |
| SSc-ILD | Systemic sclerosis associated interstitial lung disease |
| UADR | Unexpected adverse drug reaction |
| UAE | Unexpected adverse events |
| ULN | Upper limits of normal |
| VIF | Variance Inflation factor |
| WHO ATC index | World health organization anatomical therapeutic chemical index |

Effective Date: 24-Jun-2019

## STATISTICAL ANALYSIS PLAN

## **TABLE OF CONTENTS**

| ST | ATIST | ICAL ANALYSIS PLAN | 1 |
|----|--------|-------------------------------------------|----|
| SI | GNATU | URE PAGE | 2 |
| VF | ERSION | N INFORMATION (DOCUMENT REVISION HISTORY) | 4 |
| ΑĒ | BREV | TATION | 5 |
| TA | BLE C | DF CONTENTS | 6 |
| LI | ST OF | TABLES | 8 |
| 1. | STUD | OY OVERVIEW | 9 |
| | 1.1 | STUDY OBJECTIVES | 9 |
| | 1. | 1.1 Primary objective | 9 |
| | 1. | 1.2 Secondary objective | 9 |
| | 1.2 | STUDY SIZE | 9 |
| | 1.3 | MILESTONES | 9 |
| 2. | STUD | DY POPULATION | 10 |
| | 2.1 | MAIN DIAGOSIS FOR STUDY ENTRY | 10 |
| | 2.2 | INCLUSION CRITERIA | 10 |
| | 2.3 | EXCLUSION CRITERIA | 10 |
| 3. | COM | POSITION OF SUBJECTS | 11 |
| | 3.1 | SUBJECTS WHOSE CRF WAS RETRIEVED | |
| | 3.2 | SAFETY SET | 11 |
| | 3.3 | EFFECTIVENESS SET | 11 |
| | 3.4 | LONG-TERM SAFETY SET | 11 |
| | 3.5 | LONG-TERM EFFECTIVENESS SET | |
| | 3.6 | DROPOUT | 12 |
| | 3.7 | SUBJECTS OF SPECIAL INVESTIGATION | |
| 4. | GENE | ERAL ANALYSIS CONSIDERATIONS | 12 |
| | 4.1 | STATISTICAL ANALYSIS SOFTWARE | 12 |
| | 4.2 | GENERAL CONSIDERATIONS | 12 |
| 5. | DATA | HANDLING CONVENTIONS | 12 |
| | 5.1 | HANDING OF MISSING DATA | 12 |
| | 5.2 | HANDLING OF MISSING DATES | 13 |
| | 5.3 | HANDLING OF DERIVED VARIABLES | 14 |
| | 5.4 | HOW TO HANDLE DATA ERRORS AFTER DB LOCK | 15 |
| 6. | SUBJ | ECT INFORMATION | 15 |
| | 6.1 | STUDY PERIOD AND NUMBER OF SUBJECTS | 15 |

Effective Date: 24-Jun-2019

# STATISTICAL ANALYSIS PLAN

| | 6.2 | POS' | T-MARKET SURVEILLANCE TABLES | 15 |
|---|---|---|---|---|
| | 6.3 | SUB | JECT CHARACTERISTICS | 15 |
| | | 6.3.1 | Demographics | 15 |
| | | 6.3.2 | Disease information | 15 |
| | | 6.3.3 | Subjects of special investigation. | 16 |
| | | 6.3.4 | Medical history and comorbidities. | 16 |
| | | 6.3.5 | Prior and concomitant medications. | 16 |
| | 6.4 | OFE | V ADMINISTRATION STATUS | 18 |
| 7. | SAF | ETY A | NALYSES | 18 |
| | 7.1 | SUM | IMARY OF ADVERSE EVENTS | 20 |
| | 7.2 | ANA | LYSES OF ADVERSE EVENTS | 20 |
| | 7.3 | SAF | ETY ANALYSES BY FACTORS | 21 |
| | , | 7.3.1 | Univariate analysis | 21 |
| | , | 7.3.2 | Multivariable analysis | 22 |
| | 7.4 | SUM | MARY OF ADVERSE EVENTS FOR SUBJECTS OF SPECIAL INVESTIGATION | )N22 |
| | 7.5 | SUM | MARY OF ADVERSE EVENTS FOR SUBJECTS WHO ARE NOT ELIGIBLE | 23 |
| | 7.6 | SUM | IMARY OF ADVERSE EVENTS FOR LONG-TERM SAFETY SET | 23 |
| 8. | EFF | ICACY | ANALYSIS | 24 |
| | 8.1 | MAI | N OUTCOME | 24 |
| | 8.2 | OTH | ER OUTCOMES | 24 |
| | 8.3 | UNI | VARIATE ANALYSIS | 24 |
| | 8.4 | MUI | TIVARIABLE ANALYSIS | 26 |
| 9. | APP | ENDIX | · | 26 |
| | 9.1 | | ENDIX 2 | |
| | 9.2 | APP | ENDIX 3 | 26 |
| | 9.3 | APP | ENDIX 5 | 26 |
| | 9.4 | DET | AILS OF SAES LEADING TO DEATH | 27 |
| | 9.5 | DET | AILS OF SERIOUS UNEXPECTED AES | 27 |
| 10. | ROI | LE AND | RESPONSIBILITY | 27 |
| 11. | APP | LIED S | SOPS | 27 |
| 12. | APP | LIED S | SOP SDS | 27 |
| 13. | SAS | PROG | RAM CODE | 28 |
| 14. | TAE | LE SEI | LLS | 28 |



## LIST OF TABLES

| Table 1 Milestones | 9 |
|------------------------------------|----|
| Table 2 Handling of Missing Dates | 13 |
| Table 3 Derived Variables | 14 |
| Table 4 Examples of Categorization | 17 |
| Table 5 Role and Responsibility | 27 |
| Table 6 Applied SOPs | 27 |
| Table 7 Applied SOP SDs | 28 |
| Table 8 SAS program code | 28 |
| Table 9 List of Tables | 28 |



#### 1. STUDY OVERVIEW

#### 1.1 STUDY OBJECTIVES

### 1.1.1 Primary objective

The primary objective is to monitor the safety profile of Ofev in Korean patients in a routine clinical setting.

### 1.1.2 Secondary objective

The secondary objective is to monitor the effectiveness of Ofev by evaluating the change from baseline after 12 and/or 24 weeks in the FVC (mL), % predicted FVC and overall evaluation of Korean patients.

#### 1.2 STUDY SIZE

Sample size of 3,000 patients initiating Ofev, based on the requirement of the local regulatory authority (Ministry of Food and Drug Safety, MFDS). Since IPF, SSc-ILD and PF-ILD are chronic diseases it might be restrictive to collect safety and effectiveness data in short-term (12weeks) period, all patients will be enrolled for long-term (24weeks) surveillance for maintaining approved indication. Thus, all patients will be enrolled for long-term(24weeks) surveillance, basically.

Considering total surveillance size of 3,000 cases, at least 20% (600 cases) of total would be enrolled for long-term(24weeks) surveillance, even considering follow up loss in real world clinical practice.

#### 1.3 MILESTONES

MFDS sets Ofev re-examination period from 21 Oct 2016 to 20 Oct 2022. Interim report planned biannually for the initial two years and annually thereafter by Jan 2023.

**Table 1 Milestones** 

| Milestone | Planned Date |
|--------------------------|----------------------------------|
| Start of data collection | 21 Oct 2016 (HA's approval date) |
| End of data collection | 20 Oct 2022 |
| Interim report 1-1 | 20 June 2017 |
| Interim report 1-2 | 20 Dec 2017 |



| Milestone | Planned Date |
|--------------------------------|--------------|
| Interim report 2-1 | 20 June 2018 |
| Interim report 2-2 | 20 Dec 2018 |
| Third-year report | 20 Dec 2019 |
| Fourth-year report | 20 Dec 2020 |
| Fifth-year report | 20 Dec 2021 |
| Final report of study results: | 20 Jan 2023 |

#### 2. STUDY POPULATION

A total of 3,000 patients will be enrolled at approximately 60 sites by as many as 60 or more NIS physicians. To minimize the selection bias at the site level, the goal is to have participating centers reflect a balance between general hospitals which has own IRB for study. The treating physicians will mainly be internists. To minimize the selection bias, consecutive patients from each site who meet inclusion criteria will be enrolled in this study.

#### 2.1 MAIN DIAGOSIS FOR STUDY ENTRY

- Patients diagnosed with idiopathic pulmonary fibrosis
- (or) Patients diagnosed with systemic sclerosis associated interstitial lung disease
- (or) patients diagnosed with chronic fibrosing ILD with a progressive phenotype

#### 2.2 INCLUSION CRITERIA

- Patients who have been started on Ofev in accordance with the approved label in Korea
- Patients who have signed on the data release consent form

#### 2.3 EXCLUSION CRITERIA

- Patients for whom Ofev is contraindicated according to local label of Ofev
  - Patients with known hypersensitivity to Ofev, peanut or soya, or to any of the excipients
  - Women who are pregnant or nursing
  - iii. Patients with moderate (Child pugh B) and severe (Child Pugh c) hepatic impairment



#### 3. COMPOSITION OF SUBJECTS

#### 3.1 SUBJECTS WHOSE CRF WAS RETRIEVED

The Subjects whose CRF was retrieved will include those whose CRF was retrieved in the relevant year.

#### 3.2 SAFETY SET

The safety set will include all subjects who signed the data release consent form to participate in this study, took Ofev once at least, and were followed up by the physician once or more. The situations excluded from the safety set are as follows.

- Cases administered prior to the conclusion of an investigation contract
- Cases administered prior to signing the consent form
- Failure of follow-up
- Violation of efficacy effectiveness, Dosage
- Didn't take at any one time with Ofev
- Dual registration
- · Violation of Inclusion/Exclusion criteria

#### 3.3 EFFECTIVENESS SET

The effectiveness set will include safety set who were evaluated for the effectiveness including overall effectiveness evaluation. The situations excluded from the effectiveness set are as follows

- Exclusion from safety evaluation
- · Omission of effectiveness evaluation
- Overall effectiveness assessed as 'unassessable'

#### 3.4 LONG-TERM SAFETY SET

The long-term safety set will include safety set who took Ofev for more than 24 weeks and were followed up by the physician 24 weeks after the date of first Ofev administration.

#### 3.5 LONG-TERM EFFECTIVENESS SET

The long-term effectiveness set will include long-term safety set and effectiveness set who were evaluated for the effectiveness including overall effectiveness evaluation 24 weeks after the date of first Ofev administration.

c39012185-01

Effective Date: 24-Jun-2019

## STATISTICAL ANALYSIS PLAN

#### 3.6 DROPOUT

Dropout include those who signed the data release consent from to participate in this study as subject but did not meet any of the inclusion criteria, do not have any prescription record of Ofev, have prescription record but have not been followed up by the physician following prescription, and started administration prior to the signed date.

#### 3.7 SUBJECTS OF SPECIAL INVESTIGATION

The subjects of special investigation will include Pediatric population(<18y old), Geriatric population(≥65y old), Pregnant women, Lactating women, Hepatic impairment, Renal impairment.

#### 4. GENERAL ANALYSIS CONSIDERATIONS

#### 4.1 STATISTICAL ANALYSIS SOFTWARE

Statistical analyses will be performed using SAS® Version 9.4 64bit (SAS Institute, Cary, NC, USA) or higher.

#### 4.2 GENERAL CONSIDERATIONS

Continuous variables will be summarized with number of subjects, means, standard deviation (SD), median, minimum, and maximum, IQR. Categorical variables will be summarized with frequency and percentage. Unless otherwise specified, statistical tests will be performed at two-sided significance level of 5% for baseline characteristics.

P-values will be presented up to four decimal places (rounded from the 5<sup>th</sup> decimal place). The values that contain decimals such as, means, standard deviation (SD), percentages will be presented up to two decimal places (rounded up from the 3<sup>rd</sup> decimal place).

#### 5. DATA HANDLING CONVENTIONS

#### 5.1 HANDING OF MISSING DATA

All endpoints will be analyzed for OC (observed case) method. In other words, missing data is not replaced.



## 5.2 HANDLING OF MISSING DATES

If there are missing dates and are used in calculations, they will be imputed as the following:

**Table 2 Handling of Missing Dates** 

| Types of Dates | Missing | Imputation | Examples |
|---|---|---|---|
| Date of the diagnosis (IPF or SSe-ILD or PF-ILD) | MM-DD | 01-01 | Collected date: 2021-UK-UK Imputed date: 2021-01-01 |
| Prior/ Concomitant medication start date | DD | 01 | Collected date: 2021-12-UK Imputed date: 2021-12-01 |
| Prior/ Concomitant<br>medication end date | MM-DD | 12-31 | Collected date: 2021-UK-UK Imputed date: 2021-12-31 |
| | DD | Last day of the month [day] | Collected date: 2021-12-UK<br>Imputed date: 2021-12-31 |
| AE onset date | DD | Step 1. For each missing/incomplete AE onset date, an interval [INT_START, INT_END] is defined. • INT_START: Min (AE end date, 01 of the reported month) • INT_END: Min (AE end date, Last date of the reported month) | Step 1. AE end date: 2020-12-05 Collected date: 2020-11-UK interval: [2020-11-01, 2020-11-30] |
| | | Step 2. 1. Date of first Ofev administration is within the interval [INT_START, INT_END]: date of first Ofev administration | |
| | | 2. Date of first Ofev administration is before INT_START: INT_START | 2. Date of first Ofev administration:<br>2020-10-30<br>Imputed date: 2020-11-01 |
| | | 3. Date of first Ofev administration is after INT_END or missing: INT_END | Date of first Ofev administration: |



| Types of Dates | Missing | Imputation | Examples |
|---|---|---|---|
| | | | 2020-12-15 |
| | | | Imputed date: 2020-11-30 |
| AE end date | YYYY-MM-DD | Date of safety assessment | Date of safety assessment: 2020-12- |
| | | | 30 |
| | | | Collected date: UK-UK-UK |
| | | | Imputed date: 2020-12-30 |
| | MM-DD | 12-31 | Collected date: 2021-UK-UK |
| | | | Imputed date: 2021-12-31 |
| | DD | Last day of the month [day] | Collected date: 2021-05-UK |
| | | | Imputed date: 2021-05-31 |

## 5.3 HANDLING OF DERIVED VARIABLES

Derived Variables will be imputed as the following.

**Table 3 Derived Variables** 

| Variable | Derivation Method |
|---|---|
| Change from baseline | Post-baseline value – Baseline value |
| rate of change (%) | Post — baseline value — Baseline value Baseline value |
| Age group | age $\geq 18y$ old and age $< 30y$ old<br>age $\geq 30y$ old and age $< 40y$ old |
| | age $\geq 40y$ old and age $< 50y$ old<br>age $\geq 50y$ old and age $< 60y$ old<br>age $\geq 60y$ old |
| Duration of disease (years) | (Date of data release consent – Date of first diagnosis)/365.25 |
| Pediatric population | <18y old, ≥18y old |
| Geriatric population | <65 old, ≥65 old |
| Duration of AE (Days) | AE end date* – AE onset date +1 *if the end date is ongoing, then the end date will be replaced with Date of safety assessment duration will be displayed including the '≥' symbol (e.g. ≥15). If the Date of safety assessment is missing, then the end date will be replaced with Date of last visit. |
| Onset duration of AE | AE onset date – Date of first Ofev administration |



#### 5.4 HOW TO HANDLE DATA ERRORS AFTER DB LOCK

If an 'Error List After DB Lock' (SD 0314 D) document according to 'SOP 0314' Database Lock is created after DB lock, the related content is not reflected in the analysis and written in the comments.

#### 6. SUBJECT INFORMATION

#### 6.1 STUDY PERIOD AND NUMBER OF SUBJECTS

The study year and study period will be presented. The number of subjects whose CRF was retrieved, safety set, effectiveness set, long-term safety set, long-term effectiveness set by year of the study will be presented.

#### 6.2 POST-MARKET SURVEILLANCE TABLES

The study sites and study Principal Investigator will be presented. The number of subjects whose CRF was retrieved, safety set, effectiveness set, long-term safety set, long-term effectiveness set by year of the study will be presented.

#### 6.3 SUBJECT CHARACTERISTICS

Subject characteristics will be performed on safety set.

## 6.3.1 Demographics

For the following variables, the continuous variables will be summarized using number of subjects, mean, SD,

median, minimum, and maximum, IQR, and the categorical variables will be summarized using number of subjects and percentages.

- Continuous variables: Age (years), Height (cm), Weight (kg), Occupation or exposure period
- Categorical variables: Age group, Gender, Smoking status, Alcohol consumption, Occupation or exposure status

#### 6.3.2 Disease information

For the following variables, the continuous variables will be summarized using number of subjects, mean, SD,

median, minimum, and maximum, IQR, and the categorical variables will be summarized using number of subjects and percentages.

c39012185-01

## STATISTICAL ANALYSIS PLAN

- Continuous variables: Duration of disease (years)
- Categorical variables: Diagnosed disease, Allergy, Child Pugh Score Class, Family history of pulmonary fibrosis/SSc-ILD, Chest HRCT evaluation, Result of lung biopsy, Medical History, Comorbidities, Prior medication, Concomitant medication

### 6.3.3 Subjects of special investigation

The following variables will be summarized using number of subjects and percentages.

- Pediatric population (<18y old, ≥18y old)
- Geriatric population (<65 old, ≥65 old)
- Pregnant women (Yes, No)
- Lactating women (Yes, No)
- Hepatic impairment (Yes, No)
- Renal impairment (Yes, No)

#### **6.3.4** Medical history and comorbidities

Previous medical history is defined as those that are checked "1" for the question "Ongoing" under [Medical History] page of the CRF, and comorbidities are defined as those that are blanked for the same question.

Medical history and comorbidities will be summarized with number of subjects, percentages and cases. Medical history and comorbidities will be coded with Medical Dictionary for Regulatory Activities (MedDRA) version 25.0 and will be summarized with system organ class (SOC) and preferred term (PT) using number of subjects, percentages and cases.

#### 6.3.5 Prior and concomitant medications

Prior medication is defined as any medication that the subjects took before the first dose of Ofev.

Concomitant medication is defined as any medication that the subjects took on or after the first dose of Ofev. Specifically, medications will be classified as the following:

Prior medication is any medication that can be classified into any of the following categories:

- Medication start date < Date of first Ofev administration OR
- Medication end date ≤ Date of first Ofev administration



Concomitant medication is any medication that can be classified into any of the following categories:

- Medication start date ≥ Date of first Ofev administration OR
- Medication end date ≥ Date of first Ofev administration OR
- Ongoing

**Table 4 Examples of Categorization** 

| Medication start date | Medication end date | Date of first | Prior | Concomitant |
|---|---|---|---|---|
| viculcation start date | Wedication end date | Ofev administration | medication | medication |
| 2020-01-01 | 2020-01-14 | 2020-01-15 | Y | - |
| 2020-01-01 | 2020-01-15 | 2020-01-15 | Y | Y |
| 2020-01-01 | 2020-01-20 | 2020-01-15 | Y | Y |
| 2020-01-01 | Ongoing | 2020-01-15 | Y | Y |
| 2020-01-15 | 2020-01-15 | 2020-01-15 | | Y |
| 2020-01-15 | 2020-01-20 | 2020-01-15 | | Y |
| 2020-01-15 | Ongoing | 2020-01-15 | | Y |
| 2020-01-20 | 2020-01-25 | 2020-01-15 | | Y |
| 2020-01-20 | Ongoing | 2020-01-15 | | Y |

In the case of [Date of first Ofev administration = medication start date = medication end date], it is included only as the concomitant medication. If it is clearly possible to classify as Prior medication\*, it is classified only as Prior medication.

If there is a missing date, Prior/concomitant medication is classified according to [5.2 Handling of Missing Dates].

Prior and concomitant medications will be summarized with number of subjects, percentages and cases. Prior and concomitant medications will be coded using the World Health Organization Anatomical Therapeutic Chemical index (WHO ATC index) version 2022 and will be summarized with Level1(anatomical main group) and Level 5 (chemical substance) using number of subjects, percentages and cases. However, if level 5 (chemical substance) doesn't exist or 'Combinations', 'Various' then level 4 (chemical subgroup) will be used instead. (If level 5 doesn't exist then a higher level will be used.)

<sup>\* (</sup>In clinical trials comparing laparoscopic procedures, preoperative medication) lidocaine



#### 6.4 OFEV ADMINISTRATION STATUS

Total duration of administration (day), Total administered dose (mg), and Average daily dose (mg) will be summarized using number of subjects, mean, SD, median, minimum, and maximum.

If the date of last administration is missing or Ofev administration status is "continuing", then the date of last administration will be replaced with date of overall effectiveness evaluation. If the date of overall effectiveness evaluation is missing, then the date of last administration will be replaced with date of last efficacy assessment of efficacy endpoints.

Each variable is defined as follows.

- Total duration of administration (day): Date of last administration Date of first administration + 1
- Total number of days administered (day): Sum of number of days administered by timepoint (Date of last administration by timepoint - Date of first administration by timepoint + 1)
- Total administered dose (mg): Sum of administered dose by timepoint (Single dose × Frequency per Day × number of days administered by timepoint)
- Average daily dose (mg): Total administered dose (mg) / Total number of days administered (day)

#### 7. SAFETY ANALYSES

Safety analyses will be performed on Safety set.

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Adverse Drug Reaction (ADR) refers to any harmful, unintended reaction to the medicinal product of any dose at which a causal relationship with the medicinal product cannot be ruled out. In the case of voluntarily reported AEs, if the causal relationship with the medicinal

c39012185-01

## STATISTICAL ANALYSIS PLAN

product of any dose is not known, it is regarded as ADR. However, if both the reporter and the manufacturer/sponsor determine that it is not related to the medicinal product of any dose, it is excluded from ADR.

The following relationship categories will be considered as ADR:

- certain
- probable/likely
- possible
- conditional/unclassified
- unassessable/unclassifiable

Serious adverse event (SAE) is AE occurring at random doses of Ofev from this study that results in one of the following outcomes:

- Results in death
- Immediately life-threatening
- Persistent or significant disability/incapacity
- Requires patient hospitalization, Prolongs patient hospitalization
- Congenital anomaly/birth defect
- Other comparable medical criteria

Unexpected adverse event (UAE) is AE not listed in the permit.

The term Adverse Event of Special Interest (AESI) relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this study, e.g. the potential for AEs based on knowledge from other compounds in the same class.

The following are considered as AESIs:

- Hepatic injury defined by the following alterations of liver parameters:
  - 1) AST or ALT  $\geq$  3 fold ULN AND total bilirubin  $\geq$  2 fold ULN measured in the same blood draw sample
  - 2) AST or ALT  $\geq$  8 fold ULN
- Adverse events relating to gastrointestinal perforation.



Adverse events leading to discontinuation refer to a case where the action taken with trial drug due to AE is discontinued or discontinuation and reintroduction.

#### 7.1 SUMMARY OF ADVERSE EVENTS

The following types of AEs will be summarized with number and cases of AEs, incidence rate and exact 95% confidence intervals.

- Adverse event (AE)
- Adverse drug reaction (ADR)
- Serious adverse event (SAE)
- Serious adverse drug reaction (SADR)
- Unexpected adverse event (UAE)
- Unexpected adverse drug reaction (UADR)
- Adverse events of special interest (AESI)
- Adverse events leading to discontinuation
- Adverse events leading to discontinuation and reintroduction

#### 7.2 ANALYSES OF ADVERSE EVENTS

The following types of AEs will be coded with MedDRA version 25.0 and will be summarized with SOC and PT using number and cases of AEs, incidence rate. The details of SAEs will also be presented in a listing.

- AE/ADR
- SAE/SADR
- UAE/UADR
- AESI
- AE leading to discontinuation
- AE classified by Intensity
- AE classified by Outcome of the event
- AE classified by Causal Relationship
- AE classified by Action taken with Ofev
- AE classified by Therapy for the event

•

The following AEs of rare (less than 0.1%) or Occasional (less than 0.1%~5%) occurrent will be coded with MedDRA version 25.0 and will be summarized with SOC and PT using number

c39012185-01

### STATISTICAL ANALYSIS PLAN

and cases of AEs, incidence rate.

- SAE/SADR
- UAE/UADR

#### 7.3 SAFETY ANALYSES BY FACTORS

#### 7.3.1 Univariate analysis

The following categorical variables will be summarized using number of subjects, number and cases of AEs, incidence rate and 95% confidence interval. AE Occurrence will be analyzed using Pearson's chi-square test or Fisher's exact test to determine if statistically significant differences exist. (However, if [Family history of pulmonary fibrosis/SSc-ILD], [Alcohol consumption], [Occupation or exposure status], [Chest HRCT evaluation] and [Result of lung biopsy] responds with [Unknown], it is excluded from Pearson's chi-square test or Fisher's exact test.)

- Diagnosed disease (IPF, SSc-ILD, PF-ILD)
- Gender (Male, Female)
- Allergy (Yes, No)
- Child Pugh Score Class (Class A, Class B, Class C, Not Applicable)
- Family history of pulmonary fibrosis/SSc-ILD (Yes, no, Unknown)
- Smoking status (Never smoked, EX-smoker, Current smoker)
- Alcohol consumption (Never, Former, Current, Unknown)
- Occupation or exposure status (Yes, no, Unknown)
- Chest HRCT evaluation (UIP pattern, probable UIP pattern, inconsistent UIP pattern, emphysema, Normal, Unknown)
- Result of lung biopsy (UIP pattern, probable UIP pattern, possible UIP pattern, inconsistent with UIP, Normal, Unknown)
- Medical History (Yes, No)
- Comorbidities (Yes, No)
- Prior medication (Yes, No)
- Concomitant medication (Yes, No)

The following continuous variables will be summarized using number of subjects. AE Occurrence will be summarized using odds ratio and 95% confidence interval by using simple logistic regression.

c39012185-01

Effective Date: 24-Jun-2019

### STATISTICAL ANALYSIS PLAN

- Age (years)
- Height (cm)
- Weight (kg)
- Occupation or exposure period
- Duration of disease (years)
- Average daily dose (mg)

Subjects of special investigation will be summarized using number of subjects, number and cases of AEs, incidence rate and 95% confidence interval. AE Occurrence will be analyzed by using Pearson's chi-squire test or Fisher's exact test to confirm statistically significant differences.

- Pediatric population (<18y old, ≥18y old)
- Geriatric population (<65 old, ≥65 old)
- Pregnant women (Yes, No)
- Lactating women (Yes, No)
- Hepatic impairment (Yes, No)
- Renal impairment (Yes, No)

#### 7.3.2 Multivariable analysis

As a result of simple logistic regression, statistically significant variables will be summarized using odds ratio and 95% confidence interval by using multiple logistic regression. (However, Variables with the Variance Inflating Factor (VIF) exceeding 10 can be excluded from the model.) The complete case analysis will be used to handle missing values of variables in the multivariate logistic regression model.

#### 7.4 SUMMARY OF ADVERSE EVENTS FOR SUBJECTS OF SPECIAL INVESTIGATION

The following types of AEs for each subject of special investigation will be summarized with number and cases of AEs, incidence rate and exact 95% confidence intervals. The details of AEs for each subject of special investigation will also be presented in a listing.

• Adverse event (AE)



- Adverse drug reaction (ADR)
- Serious adverse event (SAE)
- Serious adverse drug reaction (SADR)
- Unexpected adverse event (UAE)
- Unexpected adverse drug reaction (UADR)
- Adverse events of special interest (AESI)
- Adverse events leading to discontinuation
- Adverse events leading to discontinuation and reintroduction

#### 7.5 SUMMARY OF ADVERSE EVENTS FOR SUBJECTS WHO ARE NOT ELIGIBLE

The following types of AEs for each subject who are not eligible will be summarized with number and cases of AEs, incidence rate and exact 95% confidence intervals. The details of AEs for each subject who are not eligible will also be presented in a listing.

- Adverse event (AE)
- Adverse drug reaction (ADR)
- Serious adverse event (SAE)
- Serious adverse drug reaction (SADR)
- Unexpected adverse event (UAE)
- Unexpected adverse drug reaction (UADR)
- Adverse events of special interest (AESI)
- Adverse events leading to discontinuation
- Adverse events leading to discontinuation and reintroduction

#### 7.6 SUMMARY OF ADVERSE EVENTS FOR LONG-TERM SAFETY SET

The following types of AEs for long-term safety set will be summarized with number and cases of AEs, incidence rate and exact 95% confidence intervals. The details of AEs for long-term safety set will also be presented in a listing.

- Adverse event (AE)
- Adverse drug reaction (ADR)
- Serious adverse event (SAE)
- Serious adverse drug reaction (SADR)
- Unexpected adverse event (UAE)
- Unexpected adverse drug reaction (UADR)



- Adverse events of special interest (AESI)
- Adverse events leading to discontinuation
- Adverse events leading to discontinuation and reintroduction

#### 8. EFFICACY ANALYSIS

Efficacy analyses will be performed on Effectiveness set.

#### 8.1 MAIN OUTCOME

For FVC (mL), the changes from baseline to 12 and 24 weeks will be summarized using number of subjects, mean, SD, median, minimum, maximum and will be compared using paired t-test depending on whether the normality assumption is met.

#### 8.2 OTHER OUTCOMES

- For % predicted of FVC, the changes from baseline to 12 and 24 weeks will be summarized using number of subjects, mean, SD, median, minimum, maximum and will be compared using paired t-test depending on whether the normality assumption is met.
- 2) For overall effectiveness evaluation, the three items ([Improved, Unchanged, Aggravated]) at the time of week 12 and week 24 will be summarized using number of subjects, percentage, 95% confidence intervals. In addition, if overall effectiveness is evaluated as [Improved], it is classified as [Efficacy]. And If overall effectiveness is evaluated as [Unchanged, Aggravated], it is classified as [Inefficacy]. [Efficacy], [Inefficacy] will be summarized using number of subjects, percentage, 95% confidence intervals. The analysis of the overall effectiveness evaluation results also will be performed on long-term effectiveness set.

#### 8.3 UNIVARIATE ANALYSIS

The following categorical variables will be summarized using number of subjects, number and cases of efficacy, efficacy rate and 95% confidence interval. Efficacy will be analyzed by using Pearson's chi-squire test or Fisher's exact test to determine if statistically significant differences exist. (However, if [Family history of pulmonary fibrosis/SSc-ILD], [Alcohol consumption], [Occupation or exposure status], [Chest HRCT evaluation] and [Result of lung biopsy] responds with [Unknown], it is excluded from Pearson's chi-squire test or Fisher's exact test.)

- Diagnosed disease (IPF, SSc-ILD, PF-ILD)
- Gender (Male, Female)
- Allergy (Yes, No)
- Child Pugh Score Class (Class A, Class B, Class C, Not Applicable)
- Family history of pulmonary fibrosis/SSc-ILD (Yes, no, Unknown)
- Smoking status (Never smoked, EX-smoker, Current smoker)
- Alcohol consumption (Never, Former, Current, Unknown)
- Occupation or exposure status (Yes, No, Unknown)
- Chest HRCT evaluation (UIP pattern, probable UIP pattern, inconsistent UIP pattern, emphysema, Normal, Unknown)
- Result of lung biopsy (UIP pattern, probable UIP pattern, possible UIP pattern, inconsistent with UIP, Normal, Unknown)
- Medical History (Yes, No)
- Comorbidities (Yes, No)
- Prior medication (Yes, No)
- Concomitant medication (Yes, No)

The following continuous variables will be summarized using number of subjects. Efficacy will be summarized using odds ratio and 95% confidence interval by using simple logistic regression.

- Age (years)
- Height (cm)
- Weight (kg)
- Occupation or exposure period
- Duration of disease (years)
- Average daily dose (mg)

Subjects of special investigation will be summarized using number of subjects, number and cases of efficacy, efficacy rate and 95% confidence interval. Efficacy will be analyzed by using Pearson's chi-square test or Fisher's exact test to determine if statistically significant differences exist.

• Pediatric population (<18y old, ≥18y old)

c39012185-01

## STATISTICAL ANALYSIS PLAN

- Geriatric population (<65y old, ≥65y old)</li>
- Pregnant women (Yes, No)
- Lactating women (Yes, No)
- Hepatic impairment (Yes, No)
- Renal impairment (Yes, No)

#### 8.4 MULTIVARIABLE ANALYSIS

As a result of simple logistic regression, statistically significant variables will be summarized using odds ratio and 95% confidence interval by using multiple logistic regression. (However, Variables with the VIF exceeding 10 can be excluded from the model.) The complete case analysis will be used to handle missing values of variables in the multivariate logistic regression model.

#### 9. APPENDIX

#### 9.1 APPENDIX 2

Appendix 2 will be prepared for the Use Result Surveillance. The number of subjects whose CRF was retrieved, safety set, effectiveness set, long-term safety set, long-term effectiveness set by year of the study will be presented. The number of subjects excluded from the safety evaluation, efficacy evaluation, long-term safety evaluation, long-term efficacy evaluation and their specific reasons will be presented.

#### 9.2 APPENDIX 3

ADR collected in use result surveillance will be summarized using number of study sites, number of safety set, number and cases of ADRs, incidence rate of ADRs according to the appendix format. AEs, SADRs, Not SAEs, Not SADRs collected from use result surveillance, special study (Pharmacoepidemiology study, etc.), clinical trials and Spontaneous reporting will be coded with Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized with system organ class (SOC) and preferred term (PT) using number and cases, incidence rate, percentage of cases (only use result surveillance).

#### 9.3 APPENDIX 5

AEs, SADRs, UADRs collected from use result surveillance, special study(Pharmacoepidemiology study, etc.), clinical trials and Spontaneous reporting will only be presented for Re-examination according to the format

#### 9.4 DETAILS OF SAES LEADING TO DEATH

The details of SAEs leading to death collected from use result surveillance, special study (Pharmacoepidemiology study, etc.), clinical trials and Spontaneous reporting will be presented in a listing.

#### 9.5 DETAILS OF SERIOUS UNEXPECTED AES

The details of Serious Unexpected AEs leading to death collected from use result surveillance, special study (Pharmacoepidemiology study, etc.), clinical trials and Spontaneous reporting will be presented in a listing.

#### 10. ROLE AND RESPONSIBILITY

Roles and responsibilities of this study are as following.

**Table 5 Role and Responsibility** 

| Role | Name | Responsibility |
|---|---|---|
| Biostatistician | | Statistical analysis |
| Senior Biostatistician | | Quality control for the statistical analysis process, Approval for SAP |

### 11. APPLIED SOPS

The following SOPs of will be applied in this study.

## **Table 6 Applied SOPs**

| SOP No. | SOP Version | SOP Name |
|---------|-------------|------------------------------------------|
| 0400 | V 3.0 | Statistical Analysis Plan |
| 0401 | V 4.1 | Statistical Analysis Process |
| 0406 | V 4.0 | Definition of Analysis Population |
| 0408 | V 3.0 | Statistical Analysis Document Management |

### 12. APPLIED SOP SDS

The following Supporting Documents of will be used in this study.



## **Table 7 Applied SOP SDs**

| SD No. | SD Version | SD Title |
|-----------|------------|-----------------------------------|
| SD 0400 A | V 3.0 | Statistical Analysis Plan |
| SD 0401 A | V 3.0 | Statistical Analysis QC Report |
| SD 0406 A | V 5.0 | Definition of Analysis Population |
| SD 0408 A | V 4.0 | STAT Master File Index |

## 13. SAS PROGRAM CODE

The following SAS program codes will be used.

Table 8 SAS program code

| Analysis method | SAS program code |
|------------------------------|--------------------------------------------|
| Pearson's chi-square test or | PROC FREQ DATA=dataset; |
| Fisher's exact test | TABLE ae*factor/CHISQ EXACT; |
| | RUN; |
| Simple logistic regression | PROC LOGISTIC DATA=dataset; |
| | CLASS factor; |
| | MODEL ae=factor; |
| | RUN; |
| Multiple logistic regression | PROC LOGISTIC DATA=dataset; |
| | CLASS factor1 factor2 factor3; |
| | MODEL ae= factor1 factor2 factor3 factor4; |
| | RUN; |

### 14. TABLE SELLS

The following are the lists of tables for this study.

**Table 9 List of Tables** 

| Table Number | Table Description |
|--------------|-------------------------------------|
| Al | Study period and number of subjects |
| A2 | Post-Market Surveillance tables |

| B1 | |
|-----|-------------------------------------------------------------------|
| | Demographics |
| B2 | Disease information |
| B3 | subjects of special investigation |
| B4 | Medical history |
| B5 | comorbidities |
| B6 | Prior medication |
| B7 | Concomitant medication |
| B8 | Ofev administration status |
| C1 | Summary of AEs |
| C2 | Status of AEs and ADRs |
| C3 | Status of SAEs and SADRs |
| C4 | Status of UAEs and UADRs |
| C5 | Status of AESI |
| C6 | Status of AEs leading to discontinuation |
| C7 | Status of AEs leading to discontinuation and reintroduction |
| C8 | Details of SAEs |
| С9 | AE classified by intensity |
| C10 | AE classified by outcome of the event |
| C11 | AE classified by causal relationship |
| C12 | AE classified by action taken with Ofev |
| C13 | AE classified by therapy for the event |
| C14 | Status of SAEs and SADRs by frequency of occurrence |
| C15 | Status of UAEs and UADRs by frequency of occurrence |
| C16 | Status of AEs by subject characteristics - categorical variables |
| C17 | Status of AEs by subject characteristics - continuous variables |
| C18 | Status of AEs for subjects of special investigation |
| C19 | Status of AEs by subject characteristics - multivariable analysis |
| C20 | Summary of AEs for subjects of special investigation |
| C21 | Details of AEs for subjects of special investigation |
| C22 | Summary of AEs for subjects who are not eligible |
| C23 | Details of AEs for subjects who are not eligible |
| C24 | Summary of AEs for Long-term Safety Set |
| C25 | Details of AEs for Long-term Safety Set |

Effective Date: 24-Jun-2019



## STATISTICAL ANALYSIS PLAN

| Table Number | Table Description |
|---|---|
| D1 | Outcome-FVC(mL) |
| D2 | Outcome – % predicted of FVC |
| D3 | Overall effectiveness evaluation |
| D4 | Result of effectiveness evaluation by subject characteristics - categorical variables |
| D5 | Result of effectiveness evaluation by subject characteristics - continuous variables |
| D6 | Effectiveness evaluation for subjects of special investigation |
| D7 | Result of effectiveness evaluation by subject characteristics - multivariable Analysis |
| D8 | Overall effectiveness evaluation for Long-term Effectiveness set |



### APPROVAL / SIGNATURE PAGE

Document Number: c39012185 Technical Version Number: 1.0

**Document Name:** 1199-0417-seap

Title: STATISTICAL ANALYSIS PLAN

## Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|-------------------------------|-----------|------------------------|
| Approval | | 30 May 2022 01:24 CEST |
| Approval-Project Statistician | | 30 May 2022 08:58 CEST |
| Approval | | 30 May 2022 16:14 CEST |
| Approval | | 03 Jun 2022 16:43 CEST |
| Approval | | 03 Jun 2022 16:47 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c39012185Technical Version Number: 1.0

(Continued) Signatures (obtained electronically)

| Meaning of Signature |
|----------------------|
|----------------------|